CLINICAL TRIAL: NCT07049939
Title: An Open-Label, Single-Dose Study to Evaluate the Effects of Hepatic Impairment on the Pharmacokinetics of MK-3543
Brief Title: A Study of Bomedemstat (MK-3543) in Participants With Mild or Moderate Hepatic Impairment (MK-3543-023)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3543-023; MK-3543-023 (Other: MSD)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — bomedemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment will receive a single oral 25 mg dose of bomedemstat on Day 1.
  Interventions: Drug: Bomedemstat
- Moderate Hepatic Impairment (Experimental): Participants with mild hepatic impairment will receive a single oral 25 mg dose of bomedemstat on Day 1.
  Interventions: Drug: Bomedemstat
- Healthy Matched Control (Experimental): Healthy participants will receive a single oral 25 mg dose of bomedemstat on Day 1.
  Interventions: Drug: Bomedemstat

INTERVENTIONS:
Drug: Bomedemstat — Capsule for oral administration
  Other Names: MK-3543

SUMMARY:
The purpose of this study is to learn what happens to bomedemstat (MK-3543) in a person's body over time. Researchers will compare what happens to bomedemstat in the body when it is given to participants with mild or moderate hepatic (liver) impairment and healthy participants.

Participants will be allocated to one of three groups: mild hepatic impairment (HI), moderate HI, or healthy matched control. All participants will receive a single oral dose of bomedemstat on Day 1.

Healthy control participants will be enrolled after hepatic impairment participants have been dosed. Healthy control participants will be matched for the mean age and mean body-mass index (BMI) of all participants with HI (mild and moderate HI combined) and sex to each HI group separately.

ELIGIBILITY:
Inclusion Criteria

The main inclusion criteria include but are not limited to the following:

* Is a non-smoker or is a moderate smoker for at least 3 months prior to dosing

Participants with Mild and Moderate HI

* Is classified as having either mild HI (Group 1) or moderate HI (Group 2) score on the Child-Pugh scale ranging from 5 to 6 (mild) or 7 to 9 (moderate)
* Has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology

Healthy Control Participants:

* Must match the mean age (± 15 years) of participants with mild HI and moderate HI
* Must match the mean body-mass index (BMI) (± 25%) of participants with mild HI (Group 1) and moderate HI
* Must match the sex ratio (±2) of participants in each HI group, separately

Exclusion Criteria

The main exclusion criteria include but are not limited to the following:

All Participants

* History of cancer (malignancy)
* Female participants of childbearing potential
* Is positive for Hepatitis C virus (HCV)
* Is positive for Hepatitis B surface antigen (HBsAg)
* Is positive for human immunodeficiency virus (HIV)

Participants with Mild and Moderate HI

* Has any significant arrhythmia or conduction abnormality
* Severe complications of liver disease within the preceding 3 months
* Primary biliary cholangitis or biliary obstruction
* Has a history of a recent variceal bleeds
* Has evidence of hepatorenal syndrome
* Has a history of liver or other solid organ transplantation
* Has an active infection requiring systemic therapy
* Requires paracentesis more often than 2 times per month
* Has transjugular intrahepatic portosystemic shunt and/or has undergone portacaval shunting

Healthy Control Participants

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is a regular user of cannabis products within approximately 6 months of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Bomedemstat in Participants with Mild Hepatic Impairment (HI) | Up to 216 hours
  Blood samples collected to determine the AUC0-inf of bomedemstat.
Maximum Plasma Concentration (Cmax) of Bomedemstat in Participants with Mild HI | Up to 216 hours
  Blood samples collected to determine the Cmax of bomedemstat.
AUC0-Inf of Bomedemstat in Participants with Moderate HI | Up to 216 hours
  Blood samples collected to determine the AUC0-inf of bomedemstat.
Cmax of Bomedemstat in Participants with Moderate HI | Up to 216 hours
  Blood samples collected to determine the Cmax of bomedemstat.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to 14 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing AEs will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to 14 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants discontinuing study treatment due to an AE will be reported.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Bomedemstat in Participants with Mild HI | Up to 216 hours
  Blood samples will be collected to determine the AUC0-last of bomedemstat.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of Bomedemstat in Participants with Mild HI | At designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24hr of bomedemstat.
Plasma Concentration at 24 Hours (C24) of Bomedemstat in Participants with Mild HI | At designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the C24 of bomedemstat.
Time to Maximum Plasma Concentration (Tmax) of Bomedemstat in Participants with Mild HI | Up to 216 hours
  Blood samples will be collected to determine the Tmax of bomedemstat.
Apparent Terminal Half-life (t1/2) of Bomedemstat in Participants with Mild HI | Up to 216 hours
  Blood samples will be collected to determine the t1/2 of bomedemstat.
Apparent Clearance (CL/F) of Bomedemstat in Participants with Mild HI | Up to 216 hours
  Blood samples will be collected to determine the CL/F of bomedemstat.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Bomedemstat in Participants with Mild HI | Up to 216 hours
  Blood samples will be collected to determine the Vz/F of bomedemstat.
AUC0-Last of Bomedemstat in Participants with Moderate HI | Up to 216 hours
  Blood samples will be collected to determine the AUC0-last of bomedemstat.
AUC0-24hrs of Bomedemstat in Participants with Moderate HI | At designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24hr of bomedemstat.
C24 of Bomedemstat in Participants with Moderate HI | At designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the C24 of bomedemstat.
Tmax of Bomedemstat in Participants with Moderate HI | Up to 216 hours
  Blood samples will be collected to determine the Tmax of bomedemstat.
t1/2 of Bomedemstat in Participants with Moderate HI | Up to 216 hours
  Blood samples will be collected to determine the t1/2 of bomedemstat.
CL/F of Bomedemstat in Participants with Moderate HI | Up to 216 hours
  Blood samples will be collected to determine the CL/F of bomedemstat.
Vz/F of Bomedemstat in Participants with Moderate HI | Up to 216 hours
  Blood samples will be collected to determine the Vz/F of bomedemstat.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - University of Miami ( Site 0003), Miami, Florida
  - Orlando Clinical Research Center ( Site 0001), Orlando, Florida
  - The Texas Liver Institute ( Site 0002), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/